CLINICAL TRIAL: NCT04556942
Title: Improvement of Cardiovascular Function After Bronchoscopic Lung Volume Reduction Using Endobronchial Valves in Patients With Severe Emphysema: A Randomized Controlled Trial
Brief Title: Improvement of Cardiovascular Function After Bronchoscopic Lung Volume Reduction Using Endobronchial Valves
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Daniel Franzen (Other)
Responsible Party: Sponsor-Investigator, Daniel Franzen, Principal Investigator, PD Dr. med. Daniel Franzen, University of Zurich
Organization: University of Zurich (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2019-01682
Record Dates: First submitted 2020-07-17; First posted 2020-09-21 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Flow Mediated Dilation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Blood Pressure; Pulse; Weights and Measures

STUDY DESIGN:
Intervention Model Description: Patients receiving routinely performed bronchoscopic lung volume reduction (BLVR) using endobronchial valves due to severe emphysema with hyperinflation are eligible for this study. After obtaining written informed consent, the participating patients will be randomized into an immediate (within 1-2 weeks) BLVR group and a delayed BLVR group (6-8 weeks) using counted and sealed envelopes. Patients in both groups will undergo baseline study specific measurements of primary and secondary endpoints (T0). The immediate BLVR group will be re-assessed 4-6 weeks after successful endobronchial valve (EBV) treatment, whereas the delayed BLVR group will be re-assessed prior EBV treatment (T1). Results of group 1 and 2 will be compared for final analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Immediate Group) (Experimental): Group 1:
  Will receive at time T0 the baseline study specific measurements of the primary and secondary endpoints:
  * Flow mediated dilation measurement
  * Blood pressure, pulse, blood oxygenation saturation measurement
  * Fit bit tracker counting steps and distance during 7 days
  * SGRQ (St Georg Respiratory Questionnaire)
  * Withdrawal of a blood sample for preservation for later examinations
  This group will receive endobronchial valve placement (EVP) within 1-2 weeks after T0.
  At T1 which will be 4-6 weeks after EVP the measurements done at T0 will be repeated.
  Interventions: Diagnostic Test: Flow Mediated Dilation (FMD) measurement; Other: Blood pressure, pulse and blood oxygen saturation measurement; Other: ST George Respiratory Questionnaire; Other: Physical activity level (PAL) measurement; Biological: Withdrawal of a blood sample; Procedure: Immediate Bronchoscopic Lung Volume Reduction
- Group 2 (Delayed Group) (Other): Group 2:
  Will receive at time T0 the baseline study specific measurements of the primary and secondary endpoints:
  * Flow mediated dilation measurement
  * Blood pressure, pulse, blood oxygenation saturation
  * Fit bit tracker counting steps and distance during 7 days
  * SGRQ (St Georg Respiratory Questionnaire)
  * Withdrawal of a blood sample for preservation for later examinations
  This group will receive endobronchial valve placement (EVP) 6-8 weeks after T0. A few days before that the investigators repeat the measurement taken at T0.
  Interventions: Diagnostic Test: Flow Mediated Dilation (FMD) measurement; Other: Blood pressure, pulse and blood oxygen saturation measurement; Other: ST George Respiratory Questionnaire; Other: Physical activity level (PAL) measurement; Biological: Withdrawal of a blood sample; Procedure: Delayed Bronchoscopic Lung Volume Reduction

INTERVENTIONS:
Diagnostic Test: Flow Mediated Dilation (FMD) measurement — FMD measurements will be performed by ultrasound using longitudinal images of the brachial artery using a high-frequency (10.0-MHz) ultrasound scanning probe (VividTM E9 with XDeclearTM; GE Healthcare, Chicago, Illinois, USA) proximal to the antecubital fossa. Two-dimensional images, acquired with electrocardiogram gating, will be obtained at baseline with Doppler ultrasound imaging to assess arterial diameter and flow velocity. Reactive hyperemia will then be induced by inflation of a pneumatic tourniquet around the forearm to at least 200 mm Hg (or > 50mmHg above systolic pressure) for 5 minutes. Post-deflation diameter and flow velocity will be monitored continuously from deflation for 210 seconds. To assess endothelial-independent vasodilation maximal brachial artery diameter will be measured continuously for 3 minutes after a single sublingual dose of nitroglycerin (NTG, 0.4 mg).
Other: Blood pressure, pulse and blood oxygen saturation measurement — Blood pressure measurement will be done with a pneumatic tourniquet on the upper arm, after at least 10 minutes rest of the patient.
  Pulse measurement and oxygen saturation measurement will be done using a finger pulseoximeter, after at least 10 minutes rest of the patient.
Other: ST George Respiratory Questionnaire — The is a validated and standardized Questionnaire designed to measure health impairment in COPD patients
Other: Physical activity level (PAL) measurement — PAL will be assessed by the number of steps and kilometers per day using a triaxial accelerometer of a multisensory activity monitor (Fitbit Alta HR; Fitbit Inc., San Francisco, CA, USA). The device is worn like a watch on the wrist. The device is worn always, except while showering or swimming.
Biological: Withdrawal of a blood sample — 5ml of blood will be withdrawn and preserved after centrifugation at -50 degrees celsius for later analysis at a yet unknown time
Procedure: Immediate Bronchoscopic Lung Volume Reduction — Bronchoscopic Lung Volume Reduction by using endobronchial valve placement Within 2 weeks after T0
  Arms: Group 1 (Immediate Group)
Procedure: Delayed Bronchoscopic Lung Volume Reduction — Bronchoscopic Lung Volume Reduction by using endobronchial valve placement Within 6-8 weeks after T0 and 3-4 days after T1
  Arms: Group 2 (Delayed Group)

SUMMARY:
There is increasing evidence showing an association between COPD and cardiovascular disease which is independent from smoking. Recently, it has been shown that FMD of the brachial artery, a surrogate marker of endothelial function, is improving after lung volume reduction surgery (LVRS) in patients with severe emphysema. Thus, hyperinflation might be an independent risk factor of atherosclerosis. Bronchoscopic lung volume reduction (BLVR) using endobronchial valves is a minimal-invasive procedure to decrease hyperinflation in patients with severe emphysema. Eventually, successful BLVR with target atelectasis may have the same effect on FMD compared to LVRS, which would underpin the association between hyperinflation and endothelial function.

Patients receiving routinely performed BLVR using endobronchial valves due to severe emphysema with hyperinflation are eligible for this study. After obtaining written informed consent, the participating patients will be randomized into an immediate (within 1-2 weeks) BLVR group and a delayed BLVR group (6-8 weeks). Patients in both groups will undergo baseline measurement of primary and secondary endpoints.

Immediate BLVR group will be re-assessed 4-6 weeks after successful EBV treatment, whereas the delayed BLVR group will be re-assessed prior EBV treatment. Results of group 1 and 2 will be compared for final analysis.

DETAILED DESCRIPTION:
Several studies were able to show an association between COPD and cardiovascular disease which is independent from smoking and other traditional cardiovascular risk factors. Although the mechanisms underlying the association between COPD and cardiovascular disease are not yet completely understood, it seems reasonable to hypothesize that COPD as a cause of hypoxemia, chronic systemic inflammation, and increased oxidative stress may be an important factor in the development and progression of atherosclerosis due to impaired endothelial function.

Endothelial function can be assessed by flow-mediated dilatation (FMD) of the brachial artery, which has been shown to provide predictive information concerning the future occurrence of cardiovascular events. Thus, assessment of FMD allows to identify patients at risk of cardiovascular events in the absence of clinically apparent vascular disease. One recent study was able to show that lung volume reduction surgery (LVRS) has a beneficial effect on endothelial function and blood pressure. They concluded that hyperinflation is a risk factor of atherosclerosis independent of cigarette smoking or others.

However, hyperinflation cannot solely be treated by LVRS but also by bronchoscopic lung volume reduction (BLVR) using endobronchial valves (EBV), coils, thermal vapour ablation, or lung sealant. The positive effects of EBV on pulmonary function, quality of life and symptoms have been shown in six randomized controlled trials. However, there is no evidence on the effect of BLVR on endothelial function. With this investigator's study, the aim is to contribute to the still limited evidence on the effects of LVR on endothelial function and to confirm the association of atherosclerosis and COPD. In addition, the investigators aim is to validate the data of the study which showed that LVRS had a beneficial effect on endothelial function, by showing similar effects after BLVR.

The investigators hypothesizes, that BLVR using endobronchial valves in patients with severe emphysema will improve endothelial function as previously shown in patients after receiving LVRS.

Patients who are study-independently planned for BLVR using endobronchial valves will be screened for study inclusion. At this time, all necessary baseline data except FMD, daily physical activity measurement and the ST George Respiratory Questionnaire (SGRQ) are already existing from routine clinical practice. Data collection will need the written informed consent of the patient on the "Patient information FMD after BLVR" after receiving further information by investigators.The investigators will explain to each participant the nature of the study, its purpose, the procedures involved, the expected duration, the potential risks and benefits and any discomfort it may entail. Each participant will be informed that the participation in the study is voluntary and that he or she may withdraw from the study at any time and that withdrawal of consent will not affect his or her subsequent medical assistance and treatment. The participant will be informed that his or her medical records may be examined by authorised individuals other than their treating physician. The formal consent of a participant, using the approved consent form, will be obtained before the participant is submitted to any study intervention. The consent form will be signed and dated by the investigator or his designee at the same time as the participant sign. A copy of the signed informed consent will be given to the study participant. The consent form will be retained as part of the study records. The informed consent process will be documented in the patient file and any discrepancy to the process described in the protocol must be explained.

The investigators start the project on the 01.04.2020 and estimate a duration of approximately two years for the recruitment of 40 eligible patients. Referring to data analysis, the investigators plan to finish the project by 31.12.2022. Patients receiving routinely performed BLVR using endobronchial valves due to severe emphysema with hyperinflation are eligible for this study. After obtaining written informed consent, the participating patients will be randomized into an immediate (within 1-2 weeks) BLVR group and a delayed BLVR group (6-8 weeks) using counted and sealed envelopes. Patients in both groups will undergo baseline study specific measurements of primary and secondary endpoints (T0) (see more detailed description under the section 'Arms and Interventions'). The immediate BLVR group will be re-assessed 4-6 weeks after successful EBV treatment, whereas the delayed BLVR group will be re-assessed prior EBV treatment (T1). Results of group 1 and 2 will be compared for final analysis.

Routine data measured before and after BLVR will be included into the study as well: Pulmonary function test, 6-Minute-Walking-Test, Laboratory.

To investigate the hypothesis, whether BLVR can improve endothelial function assessed by FMD, differences in the outcomes between the group experiencing atelectasis after BLVR and the groups not experiencing atelectasis or not receiving ELVR will be evaluated by unpaired t-tests or by non-parametrical tests as appropriate. The confidence interval (CI) for statistical significance will be defined as 95%. A p value of less than .05 will be considered statistically significant. All statistical analyses will be performed by SPSS Statistics for Windows 25 (IBM, Armonk, NY). Data will be reported as median interquartile range (IQR) or as percentages, as appropriate.

The sample size was estimated on the assumption that a clinically relevant mean (SD) difference in FMD between the intervention group and the control group is 2.9% (2.1-3.6% [95% CI]) [8]. To achieve a power of 80%, 38 patients would be required to complete the study. Because of an anticipated dropout rate of two patients, 40 patients will be included.

Individual participants will not be identifiable from the results as submitted for publication. Data analysis will only use coded data records. As set out in the Informed Consent, authorized staff of the responsible Ethics Committee may obtain access to all study data under strict adherence to confidentiality rules. Patient baseline data (age, sex, BMI, smoker status, medication list), 6-minute walk test, bronchoscopy reports, lung function data, and radiological findings as well as blood pressure and heart rate measurements, lab results (CRP, BNP) and the result of the transthoracic echocardiography will be drawn from patient record files, coded and stored in hardcopy form. Where copies of the original source document as well as printouts of original electronic source documents are retained, these shall be signed and dated by a member of the investigation site team for validation of the original information. After the measurement of PAL, data will be downloaded from the Fitbit® device and stored as coded data. Data will not be accessible to the device producer and will be deleted from the device once it is transferred. Where copies of the original source document as well as printouts of original electronic source documents are retained, these shall be signed and dated by a member of the investigation site team for validation of the original information. At a later stage, pseudonym data will be analysed using statistic software (e.g. SPSS).The investigators will be responsible for data collection, confidentiality, and data management.

Data generation, transmission, archiving, and analysis of health related personal data within this project strictly follow the current Swiss legal requirements for data protection and according to ClinO, Art. 18. Prerequisite is the voluntary approval of the participant given by signing the informed consent prior start of participation of the research project.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject between 40 and 75 years of age
* Written informed consent after participant's information signed by patient
* Scheduled for BLVR using endobronchial valves at the University Hospital Zurich
* Dyspnoea at rest or at minimal physical activity (MRC score ≥2), severe limitation of exercise capacity (6-min walk distance < 500 m).
* COPD (GOLD guidelines) with severe obstructive ventilator defect (FEV1 <40% predicted)
* Functional aspects of lung emphysema with irreversible hyperinflation, defined as a residual volume to total lung capacity ratio (RV/TLC) of >0.6
* Pulmonary emphysema confirmed by high resolution computer tomography

Exclusion Criteria:

* Age < 40 years, age > 75 years
* COPD exacerbation within the last 6 weeks or > 2 exacerbations per year
* Pregnancy
* Lacking ability to form an informed consent (including impaired judgement, communication barriers)
* Current smokers
* Overt active coronary artery disease, left ventricular function impairment
* Pulmonary hypertension with a mean pulmonary artery pressure >35 mmHg at rest
* Acute bronchopulmonary infection, bronchiectasis on high resolution tomography
* Pulmonary cachexia (body mass index <18kg/m2)
* Malignant disease with a life expectancy of less than 2 years
* Addiction to alcohol/drugs (= inability to withhold intake during 1 week)

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-06-05 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Postinterventional change in endothelial function assessed by flow mediated dilation (FMD) (%) before and after the bronchoscopic lung volume reduction (BLVR). | FMD measurement will be done at baseline and once again within 6-8 weeks afterwards.
  FMD will be performed by ultrasound using longitudinal images of the brachial artery proximal to the antecubital fossa. Two-dimensional images will be obtained at baseline with Doppler ultrasound imaging to assess arterial diameter and flow velocity. Reactive hyperemia will then be induced by inflation of a pneumatic tourniquet around the forearm to at least 200 mm Hg for 5 minutes. Post-deflation diameter and flow velocity will be monitored continuously from deflation for 210 seconds. To assess endothelial-independent vasodilation maximal brachial artery diameter will be measured continuously for 3 minutes after a single sublingual dose of nitroglycerin (NTG, 0.4 mg). Brachial artery diameter will be measured automatically at the onset of the R wave with dedicated software. Results of endothelial-dependent (FMD) and endothelial-independent (NTG) vasodilation will be expressed as percent change in arterial diameter from the baseline diameter

SECONDARY OUTCOMES:
Physical activity level (PAL) measuring the steps per day, converting that into a distance in kilometers per day | Measurement at baseline and once again within 6-8 weeks afterwards.
  PAL will be assessed by the measurement of the number of steps per day. The device will calculate from the number of steps per day the distance in kilometers per day knowing the height of the patient. The height will be programmed into the device beforehand.
  To measure the steps per day the investigator uses a triaxial accelerometer of a multisensory activity monitor (Fitbit Alta HR; Fitbit Inc., San Francisco, CA, USA). The device is worn like a watch on the wrist of the patient. The device is worn always, except while showering or swimming. At both visits patients will receive the device and wear it for seven days for data collection and send it back via postal mail afterwards.
Blood pressure (mmHg) | Measurement at baseline and once again within 6-8 weeks afterwards.
  Measurement of the systolic and diastolic blood pressure is done after 10 minutes of rest using a pneumatic tourniquet and a pulseoximeter.
Heart rate (beats per minute) | Measurement at baseline and once again within 6-8 weeks afterwards.
  Measurement is done after 10 minutes of rest using a pulseoximeter.
Blood oxygen saturation (%) | Measurement at baseline and once again within 6-8 weeks afterwards.
  Measurement is done after 10 minutes of rest using a pulseoximeter.
St. George Respiratory Questionnaire (SGRQ) | Measurement at baseline and once again within 6-8 weeks afterwards.
  Standardized questionaire to assess the health impaired through COPD. It is in two parts. Part I produces the Symptoms score, and Part 2 the Activity and Impacts scores. A Total score is also produced. An excel-based scoring calculator is used to analyze the collected data. All positive responses are entered as 1 and all negative responses are entered as 0.
  Three component scores are calculated for the SGRQ:
  * Symptoms: this component is concerned with the effect of respiratory symptoms, their frequency and severity.
  * Activity: concerned with activities that cause or are limited by breathlessness
  * Impacts: covers a range of aspects concerned with social functioning and psychological disturbances resulting from airways disease A Total score is also calculated which summarises the impact of the disease on overall health status. Scores are expressed as a percentage of overall impairment where 100 represents worst possible health status and 0 indicates best possible health status.
6-minute walking distance (6-MWD) in meters | Done during the routine visit before BLVR, which is before the study phase and it will be repeated during the routine follow-up 4-6 weeks after BLVR
  This assessment is not study specific. It is done during the regular assessment before BLVR and repeated after BLVR. It measures the distance a patient can go within 6 minutes.
Forced Expiratory Volume in first second (FEV1) in liters | Done during the routine visit before BLVR, which is before the study phase and it will be repeated during the routine follow-up 4-6 weeks after BLVR
  This assessment is not study specific. It is done during the regular assessment before BLVR and repeated after BLVR. It measures the volume in liters that is exhaled during the first second of forced exhalation during a pulmonary function test.
Residual Volume (RV) in liters | Done during the routine visit before BLVR, which is before the study phase and it will be repeated during the routine follow-up 4-6 weeks after BLVR
  This assessment is not study specific. It is done during the regular assessment before BLVR and repeated after BLVR. During a pulmonary function test it measures the volume in liters that remains in the lungs after maximal exhalation .
Residual Volume (RV)/ Total Lung Capacity (TLC) in percentage | Done during the routine visit before BLVR, which is before the study phase and it will be repeated during the routine follow-up 4-6 weeks after BLVR
  This assessment is not study specific. It is done during the regular assessment before BLVR and repeated after BLVR. During a pulmonary function test it measures the Residual Volume to Total Lung Capacity Ratio expressed as percentage.
CO-Diffusion Capacity (DLCO) in percentage | Done during the routine visit before BLVR, which is before the study phase and it will be repeated during the routine follow-up 4-6 weeks after BLVR
  This assessment is not study specific. It is done during the regular assessment before BLVR and repeated after BLVR. It measures the transfer of gas from air in the lung, to the red blood cells in lung blood vessels. It is part of a comprehensive series of pulmonary function tests to determine the overall ability of the lung to transport gas into and out of the blood.
Number of participants with relevant change in C-reactive protein before and after BLVR | Done during the routine visit before BLVR, which is before the study phase and it will be repeated during the routine follow-up 4-6 weeks after BLVR
  This assessment is not study specific. In the blood C-reactive protein will be measured. It is done during the regular assessment before BLVR and repeated after BLVR. The investigator will observe if the value changes before and after the intervention.
Number of participants with relevant change NT-proBNP before and after BLVR | Done during the routine visit before BLVR, which before is the study phase and it will be repeated during the routine follow-up 4-6 weeks after BLVR
  This assessment is not study specific. In the blood NT-pro-BNP will be measured. It is done during the regular assessment before BLVR and repeated after BLVR. The investigator will observe if the value changes before and after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Franzen, PD Dr. med., Principal Investigator — Universitiy Hospital Zuich, Department of pulmonology
Locations (1):
- University Hospital Zurich, Department of Pulmonology, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Projections of global mortality and burden of disease from 2002 to 2030 — http://pubmed.ncbi.nlm.nih.gov/17132052/
- See also: Global Strategy for the Diagnosis, Management, and Prevention of Chronic Obstructive Lung Disease 2017 Report. GOLD Executive Summary — http://pubmed.ncbi.nlm.nih.gov/28128970/
- See also: Ascertainment of cause-specific mortality in COPD: operations of the TORCH Clinical Endpoint Committee — http://pubmed.ncbi.nlm.nih.gov/17311843/
- See also: Population-based study of lung function and incidence of heart failure hospitalisations — http://pubmed.ncbi.nlm.nih.gov/20627923/
- See also: The relationship between reduced lung function and cardiovascular mortality: a population-based study and a systematic review of the literature — http://pubmed.ncbi.nlm.nih.gov/15947307/
- See also: Cardiovascular disease in patients with chronic obstructive pulmonary disease, Saskatchewan Canada cardiovascular disease in COPD patients — http://pubmed.ncbi.nlm.nih.gov/16039877/
- See also: Hospitalizations and mortality in the Lung Health Study — http://pubmed.ncbi.nlm.nih.gov/12153966/
- See also: Lung Volume Reduction Surgery and Improvement of Endothelial Function and Blood Pressure in Patients with Chronic Obstructive Pulmonary Disease. A Randomized Controlled Trial — http://pubmed.ncbi.nlm.nih.gov/26016823/
- See also: Raised CRP levels mark metabolic and functional impairment in advanced COPD — http://pubmed.ncbi.nlm.nih.gov/16055618/
- See also: C-reactive protein and mortality in mild to moderate chronic obstructive pulmonary disease — http://pubmed.ncbi.nlm.nih.gov/16738034/
- See also: Effects of oxygen on autonomic nervous system dysfunction in patients with chronic obstructive pulmonary disease — http://pubmed.ncbi.nlm.nih.gov/10836335/
- See also: Pulmonary and systemic oxidant/antioxidant imbalance in chronic obstructive pulmonary disease — http://pubmed.ncbi.nlm.nih.gov/16113469/
- See also: Arterial Stiffness Is Independently Associated with Emphysema Severity in Patients with Chronic Obstructive Pulmonary Disease — http://www.atsjournals.org/doi/full/10.1164/rccm.200707-1080OC
- See also: Determinants of systemic vascular function in patients with stable chronic obstructive pulmonary disease — http://pubmed.ncbi.nlm.nih.gov/18836149/
- See also: Assessment of endothelial function by non-invasive peripheral arterial tonometry predicts late cardiovascular adverse events — http://pubmed.ncbi.nlm.nih.gov/20181680/
- See also: Non-invasive detection of endothelial dysfunction in children and adults at risk of atherosclerosis — http://pubmed.ncbi.nlm.nih.gov/1359209/
- See also: Risk stratification for postoperative cardiovascular events via noninvasive assessment of endothelial function: a prospective study — http://pubmed.ncbi.nlm.nih.gov/11927524/
- See also: Surgical and endoscopic interventions that reduce lung volume for emphysema: a systemic review and meta-analysis — http://pubmed.ncbi.nlm.nih.gov/30744937/
- See also: Expert consensus and evidence-based recommendations for the assessment of flow-mediated dilation in humans — http://pubmed.ncbi.nlm.nih.gov/31211361/